CLINICAL TRIAL: NCT01584622
Title: Clinical Evaluation of the CADence System in Detection of Coronary Artery Diseases
Brief Title: Clinical Evaluation of the CADenceTM System in Detection of Coronary Artery Diseases
Acronym: CADENCE
Status: Withdrawn | Phase: Not Applicable | Type: Interventional
Sponsor: AUM Cardiovascular, Inc. (Industry)
Responsible Party: Sponsor
Allocation: Not Applicable | Model: Single Group | Masking: Double | Purpose: Diagnostic
Other Study IDs: AUM1040-001
Record Dates: First submitted 2012-04-02; First posted 2012-04-25 (Estimated); Last update posted 2013-07-01 (Estimated); Status verified 2013-06

CONDITIONS: Coronary Artery Disease
MeSH Terms: conditions — Coronary Artery Disease

STUDY DESIGN:
Who Masked: Investigator, Outcomes Assessor
Oversight: Data Monitoring Committee: No

INTERVENTIONS:
Device: CADence System — Non-invasive detection of > or equal to 50% stenosis in any of the major coronary arteries.
  Other Names: AUM Cardiovascular, Inc.

SUMMARY:
The purpose of the study is to evaluate the effectiveness of the CADence system, a non-invasive device, in detecting greater than or equal to 50% coronary stenosis anywhere in the coronary tree.

ELIGIBILITY:
Inclusion Criteria:

* Over 18 years old
* Willing and able to give informed consent
* Indicated for angiography evaluation.

Exclusion Criteria:

* Pregnant or nursing
* Presence of pacemaker/defibrillator
* Presence of artificial valve
* Presence of severe valve disease
* Presence of congenital heart defect
* Left Ventricular Assist Device (LVAD)
* Presence of a bypass graft
* Presence of scars on the site thorax areas
* Coarctation of the aorta
* Participation in trial within 30 days prior to collecting CADenceTM data
* Asthma with wheezing
* Inability to lie flat in the supine position
* Acute STEMI
* Heart Transplant
* Recent Cocaine Use

Min Age: 18 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 0 (Actual)
Dates: Start 2012-07; Primary Completion 2012-12 (Estimated); Study Completion 2013-02 (Estimated)

PRIMARY OUTCOMES:
Efficacy of CADence in detecting greater than or equal to 50% stenosis anywhere in the coronary tree. | within three months
  The CADence System will be considered to have demonstrated effectiveness in detecting greater than or equal to 50% coronary artery stenosis anywhere in the coronary tree if the estimated sensitivity as compared to angiography is statistically higher than 70%.

CONTACTS AND LOCATIONS:
Overall Officials: Robert Wilson, MD, Study Chair — University of Minnesota; Roxana Mehran, MD, Study Chair — Mt. Sinai; James Chapman, MD, Principal Investigator — Cheyenne Vascular & Heart Institute; Mark Tannenbaum, PhD, Principal Investigator — Iowa Heart Center; Robert Schwartz, MD, Principal Investigator — Abbott/Minneapolis Heart Institute; Jeff Chambers, MD, Principal Investigator — Mercy Hospital; Giora Weisz, MD, Principal Investigator — Columbia University
Locations (7):
- United States (7):
  - Iowa Heart Center, Des Moines, Iowa
  - Mercy Hospital, Coon Rapids, Minnesota
  - Abbott/Minneapolis Heart Institute, Minneapolis, Minnesota
  - University of Minnesota, Minneapolis, Minnesota
  - Columbia University, New York, New York
  - Mt. Sinai, New York, New York
  - Cheyenne Vascular & Heart Institute, Cheyenne, Wyoming